CLINICAL TRIAL: NCT06051383
Title: Building Patient Capability for Managing Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amna A. Desouky, MD (Other)
Responsible Party: Sponsor-Investigator, Amna A. Desouky, MD, Assistant Professor of Medical Surgical Nursing, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Self-management
Record Dates: First submitted 2023-09-18; First posted 2023-09-22 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Self-Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Experimental): Research design:
  Quasi-experimental, single group pre- posttest design was utilized in the study. all patients will be assessed for LUTS at base line then will be reassessed after three months.
  Study variables:
  The independent variable is self management intervention while the dependent variable is the severity of lower urinary tract symptoms.
  Interventions: Other: Self management

INTERVENTIONS:
Other: Self management — patients will be assessed at base line using tool I,II Patients will receive self-management intervention in the form of sessions. Four to six patients in each session. Each session will last approximately 20 minutes
  Session 1 :
  * Introduction to the concept of self-management.
  * Education/reassurance
  * Managing fluid intake.
  * Caffeine abstinence
  * Alcohol advice
  Session 2 :
  * Adjusting medications
  * Constipation advice.
  * Strategies for dribbling. pelvic floor exercise.
  * Double-voiding.
  * Bladder re-training.
  Session 3:
  • Booster session All sessions are supported with a self-management booklet given in session. All patients will be reassessed after three months

SUMMARY:
Aim of this study is to evaluate the effect of conducting self-management interventions on severity of lower urinary tract symptoms (LUTS) for patients with benign prostatic hyperplasia (BPH).

Research hypothesis:

To fulfill the aim of this study, the following research hypothesis was formulated:

Patients with benign prostatic hyperplasia will suffer less lower urinary tract symptoms (LUTS) after conducting self-management intervention than before conducting.

DETAILED DESCRIPTION:
Research design: Quasi-experimental (pre-posttest) research design was utilized to conduct this study.

This study was conducted at Assiut Urology and Nephrology Hospital. A purposive sample of 60 adult male patients diagnosed with benign prostatic hyperplasia were older than 40 years old, had no other factors influencing their urination, such as prostate cancer.

Patients had been assessed at base line using the following tools:

Tool (I): A structured interview questionnaire. Tool (II): International Prostate Symptom Score (IPSS).

Each patient will be assessed before conducting self-management intervention for socio-demographic data, clinical data, and patients' knowledge regarding self-management using the tool I.

Each patient will be assessed for lower urinary tract symptoms before conducting self-management intervention using tool tool II(IPSS).

IPSS is a scoring system used to screen for and diagnose BPH as well as to monitor symptoms and guide decisions about how to manage the disease monitor lower urinary tract symptoms, It includes seven questions, about symptom of BPH.Each question had a range from 0 to 5 for its answer. Maximum score of 35 points. On the basis of total score, the symptoms were categorized into mild (0 -7), moderate (8-19), and severe (20-35).

After 3 months from conducting self-management intervention each patient was reassessed for clinical progression "severity" of lower urinary tract symptoms(LUTS)using (tools II).

ELIGIBILITY:
Inclusion:

* Adult patients.
* Men.
* Clinical diagnosis of benign prostatic hyperplasia.

Exclusion:

* Prostate cancer.
* Severe symptoms necessitating surgical treatment.
* Uncontrolled diabetes.
* End-stage cardiac disease or respiratory failure.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients diagnosed with benign prostatic hyperplasia
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Severity of lower urinary tract symptoms of benign prostate hyperplasia. | Three months
  Evaluate outcome of conducting self-management intervention sessions on clinical progression of lower urinary tract symptoms of benign prostate hyperplasia.
  through assessing
  Lower urinary tract symptoms of benign prostate hyperplasia before and after self-management intervention by using international prostate symptom score (IPSS)
  The IPSS was developed by American Urological Association, 1992. Is a scoring system used to screen for and diagnose BPH as well as to monitor symptoms and guide decisions about how to manage the disease, It includes seven questions, about symptom of BPH that asked to the patients about how often they have. Each question had a range 5 from 0 to 5 for its answer. Maximum score of 35 points. On the basis of total score, the symptoms were categorized into mild (0 -7), moderate (8-19), and severe (20-35).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No